CLINICAL TRIAL: NCT03005795
Title: Does Mozart Reduces Anxiety in Women With Cervical Dysplasia? A Randomized Controlled Trial.
Brief Title: Music and Colposcopy in Women With Cervical Dysplasia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zydolab - Institute of Cytology and Immune Cytochemistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: COLPO-3
Record Dates: First submitted 2016-12-25; First posted 2016-12-29 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Uterine Cervical Dysplasia
Keywords: cervical dysplasia; colposcopy; anxiety; music; mozart; randomized controlled trial
MeSH Terms: conditions — Uterine Cervical Dysplasia; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music and colposcopy (Experimental): Women will hear Mozarts symphony Nr. 40 during the colposcopic examination
  Interventions: Device: Headphones
- Colposcopy without music (Active Comparator): During the colposcopic examination women will not hear music
  Interventions: Other: No Headphones

INTERVENTIONS:
Device: Headphones — Music can be heard through headphones
  Arms: Music and colposcopy
Other: No Headphones — No Headphones will be used.
  Arms: Colposcopy without music

SUMMARY:
To assess the effect of music during colposcopy on women´s anxiety.

ELIGIBILITY:
Inclusion Criteria:

* women referred for colposcopy due to cervical abnormalities
* We included women if they attended colposcopy for the first time

Exclusion Criteria:

* pregnant women
* presence of a language barrier
* known anxiety disorder or depression
* history of conization or other treatments on the cervix uteri
* known oncological disorder
* auditory defect
* cardiovascular disease
* inadequate colposcopy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-07 (Actual)

PRIMARY OUTCOMES:
Change in anxiety scores | 10 minutes before and after colposcopy
  Each women completes the state anxiety questionnaire (state-trait anxiety inventory [STAI]) 10 minutes before and 10 minutes after colposcopy. The difference in scores before and after colposcopy will be measured.

SECONDARY OUTCOMES:
Anxiety score after colposcopy | 10 minutes before and after colposcopy
  Each women completes the state anxiety questionnaire (state-trait anxiety inventory [STAI]) 10 minutes after colposcopy.
Change in heart rate | 10 minutes
  The difference in heart rate before and after colposcopy will be measured.
Pain during examination | 10 minutes
  women scores their pain level using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 (,no pain') to 10 (,worst imaginable pain').
Pain after examination | 10 minutes
  women scores their pain level using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 (,no pain') to 10 (,worst imaginable pain').
general unpleasantness during examination | 10 minutes
  women scores their feeeling during colposcopy using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 ("not at all unpleasant") to 10 ("extremely unpleasant").
Anxiety during examination | 10 minutes
  women scores their anxiety during colposcopy using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 ("no anxiety at all") to 10 ("worst imaginable anxiety")
Overall Satisfaction | 10 minutes
  women scores their satisfaction using a horizontal 100-mm visual analogue scale (VAS) ranging from 0 ("maximally unsatisfied") to 10 ("maximally satisfied").

CONTACTS AND LOCATIONS:
Overall Officials: Ziad Hilal, M.D., Principal Investigator — Zydolab - Institute of Cytology and Immune Cytochemistry
Locations (2):
- Germany (2):
  - Zydolab - Institute of Cytology and Immune Cytochemistry, Dortmund, North Rhine-Westphalia
  - Department of Obstetrics and Gynecology of the Ruhr University Bochum, Herne, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hilal Z, Alici F, Tempfer CB, Rath K, Nar K, Rezniczek GA. Mozart for Reducing Patient Anxiety During Colposcopy: A Randomized Controlled Trial. Obstet Gynecol. 2018 Oct;132(4):1047-1055. doi: 10.1097/AOG.0000000000002876. PMID 30204685